CLINICAL TRIAL: NCT00206102
Title: A Multicenter, Open Label, Flexible-dose, Parallel-group Evaluation of the Cataractogenic Potential of Quetiapine Fumarate (Seroquel) and Risperidone (Risperdal) in the Long Term Treatment of Participants With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of the Cataractogenic Potential of Seroquel and Risperdal in the Treatment of Participants With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5077IL/0089; D1441C00089
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate; Risperidone

ARMS (2):
- 1 (Experimental): Quetiapine fumarate
  Interventions: Drug: quetiapine fumarate
- 2 (Active Comparator): Risperidone
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: quetiapine fumarate — flexible dose oral
  Other Names: Seroquel; ICI 204,636
  Arms: 1
Drug: risperidone — flexible dose oral
  Arms: 2

SUMMARY:
This Phase IV, randomized, parallel-group study is designed to evaluate the cataractogenic potential of quetiapine fumarate (SEROQUEL) compared with that of a putative non-cataractogenic antipsychotic medication risperidone (RISPERDAL). This study is being conducted to fulfill the SEROQUEL Phase IV commitment regarding evaluation of cataractogenic potential.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 65
* Both Eyes present with lenses intact (no previous cataract extractions)
* Stable place of residency

Exclusion Criteria:

* History of corneal surgery
* Legal blindness (defined as best corrected visual acuity of 20/200 or worse in one or both eyes
* Previous participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1098 (Actual)
Dates: Start 2003-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (63):
- United States (63):
  - Research Site, Little Rock, Arkansas
  - Research Site, Mabelvale, Arkansas
  - Research Site, Morrilton, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Chula Vista, California
  - Research Site, Garden Grove, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, San Marcos, California
  - Research Site, Denver, Colorado
  - Research Site, New Britian, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Oak Brook Terrace, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Stratford, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Beechwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Medina, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Media, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Midvale, Utah
  - Research Site, Arlington, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 24-month, multi-center, evaluator masked (ophthalmologist), open-label, flexible-dose, parallel-group study, 82 sites recruited Sept 2003 through Oct 2008. In total 1099 participants were randomized by Interactive Voice Response System (IVRS). One excluded participant was randomized before the rand visit, and never returned to any study visits.
Pre-assignment Details: Screening for eligibility and must be cross-tapered off of all previous antipsychotic medications
Groups:
- Quetiapine Fumarate: Quetiapine fumarate - flexibly dosed (200 - 800 mg/day)
- Risperidone: Risperidone - flexibly dosed (2 - 8 mg/day)
Period: Overall Study
Arm/Group | Quetiapine Fumarate | Risperidone
Started | 596 | 502
Completed | 188 | 187
Not Completed | 408 | 315
Not completed — Adverse Event | 119 | 82
Not completed — Protocol Violation | 0 | 2
Not completed — Lack of therapeutic response | 16 | 11
Not completed — Lost to Follow-up | 95 | 66
Not completed — Withdrawal by Subject | 118 | 101
Not completed — Study-specific discontinuation criteria | 18 | 17
Not completed — None of those categories | 42 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine Fumarate | Risperidone | Total
Number analyzed (Participants) | 596 | 502 | 1098
Age, Customized [Number; unit: Participants]
  < 40 years | 265 | 223 | 488
  40 to 65 years | 331 | 279 | 610
Sex: Female, Male [Count of Participants; unit: Participants] — Participants in the United States (USA) randomized by the study's Interactive Voice Response System (IVRS).
  Participants
    Female | 253 | 199 | 452
    Male | 343 | 303 | 646

OUTCOME MEASURES:

1. Primary Outcome: Presence of a Cortical (C) Type of Cataractogenic Potential Events in Participants as Assessed and Agreed by 2 Independent, Treatment-masked Ophthalmologists Using the Lens Opacities Classification System II (LOCS II ) Grading Scale
Description: Presence of C type of cataractogenic potential event in participant was defined if any LOCS II grades of 2, 3, 4, 5 (with any grade of 0, trace,1 at randomization) assessed and agreed by 2 independent, treatment-masked ophthalmologists at any post-randomization assessment in one or both eyes. 0= no cataract; 5 is worst. There are no subscales. 0 is the best, 5 is the worst.
Time Frame: Randomization to Month 24
Population: The 2-year eye per protocol (E2PP) analysis included all randomized participants who met eye eligibility, had a valid baseline LOCS II evaluation, had reached the study endpoint of either a LOCS II identified cataractogenic potential event or dosed for 21 months without a LOCS II event, and had no major protocol deviations.
Measure: Number; unit: Participants with C type event
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 161 | 168
Participants with C type event | 2 | 8

2. Primary Outcome: Presence of a Nuclear Opalescence (N) Type of Cataractogenic Potential Events in Participants as Assessed and Agreed by 2 Independent, Treatment-masked Ophthalmologists Using the LOCS II Grading Scale
Description: Presence of N type of cataractogenic potential event in Participants was defined if any LOCS II grades of 2, 3, 4 (with grade at rand equals 0,1), or if the LOCS II grades of 3,or 4 (with grade at randomization=2) assessed and agreed by 2 independent, treatment-masked ophthalmologists at any post-randomization assessment in one or both eyes. 0 is the best, 4 is the worst.
Time Frame: Randomization to Month 24
Population: as for outcome 1
Measure: Number; unit: Participants with N type event
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 161 | 168
Participants with N type event | 0 | 2

3. Primary Outcome: Presence of a Posterior Subcapsular (P) Type Cataractogenic Potential Events in Participants as Assessed and Agreed by 2 Independent, Treatment-masked Ophthalmologists Using the LOCS II Grading Scale
Description: Presence of P type of cataractogenic potential event in participant was defined if any LOCS II grades of 1, 2, 3 , 4 (with grade=0 at randomization) assessed and agreed by 2 independent, treatment-masked ophthalmologists at any post-randomization assessment in one or both eyes. 0 is the best, 4 is the worst.
Time Frame: Randomization to Month 24
Population: as for outcome 1
Measure: Number; unit: Participants with P type event
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 161 | 168
Participants with P type event | 4 | 7

4. Secondary Outcome: Change in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS total score equals sum of the 30-items scores (range: 30-210). Each item has ( 1-7 units), 1 indicates "absent" psychosis symptom, and 7 - "extreme" symptom degree. Change in PANSS total score : total score at month 24 minus total score at randomization.Alleviation of psychotic symptoms are indicated by a negative change in PANSS total score.
Time Frame: Randomization to Month 24
Population: The intention-to-treat for psychiatric assessments (ITTP) analysis included all randomized participants who had a valid baseline and at least 1 post baseline assessment of PANSS total score, and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | -9.1 (15.4) | -8.6 (16.6)

5. Secondary Outcome: Change in the PANSS Positive Subscale Score
Description: PANSS Positive subscale score equals sum of the 7-items scores(range:7-49). Each item has ( 1-7 units), 1 indicates "absent" psychosis symptom, and 7 - "extreme" symptom degree.
Time Frame: Randomization to Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | -2.7 (5.3) | -2.8 (5.1)

6. Secondary Outcome: Change in the PANSS Negative Subscale Score
Description: PANSS Negative subscale score equals sum of the 7-items scores(range:7-49). Each item has ( 1-7 units), 1 indicates "absent" psychosis symptom, and 7 - "extreme" symptom degree. Change in PANSS Negative subscale score:score at month 24 minus score at randomization. Alleviation of negative psychotic symptoms are indicated by a negative change score.
Time Frame: Randomization to Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | -2.2 (5.5) | -1.5 (5.7)

7. Secondary Outcome: Change in the PANSS Psychopathology Subscale Score
Description: PANSS psychopathology subscale score equals sum of the 16-items scores(range:16-112). Each item has ( 1-7 units),1= "absent" psychosis symptom, 7= "extreme" symptom degree.Change in PANSS psychopathology subscale:score at month 24 minus score at randomization. Alleviation of general psychopathology symptoms are indicated by a negative change score.
Time Frame: Randomization to Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 161 | 168
units on scale | -4.2 (7.7) | -4.4 (8.8)

8. Secondary Outcome: Change in the Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: CGI-S score is accessed on a seven-graded scale ranging from most extremely ill/ very much worse (7) to normal/very much improved (1) , 1 is best. Change : score at month 24 minus score at randomization.
Time Frame: Randomization to Month 24
Population: The intention-to-treat for psychiatric assessments (ITTP) analysis included all randomized participants who had a valid baseline and at least 1 post baseline assessment of PANSS total score (not related to CGI-S), and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | -0.7 (0.9) | -0.5 (1.0)

9. Secondary Outcome: Change in Health-related Quality of Life as Measured by Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q SF) Total Score
Description: Q-LES-Q total score is the sum of the 16 times of Q-LES-Q SF(range:16-80).Each item has a 5 point satisfaction level scale:from 1=very poor(worst value) to 5=very good(best).Larger values indicate a higher perceived quality of life enjoyment and satisfaction.Change in Q-LES-Q total score:total score at month 24 minus total score at randomization
Time Frame: Randomization to Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | 2.4 (11.6) | 2.7 (10.4)

10. Secondary Outcome: Change in Personal Evaluation of Transitions in Treatment (PETiT) Total Score
Description: PETiT total score is the sum of the 30 items of PETiT questionnaire(range:0-60) on subjects perceived well-being, adherence, tolerability, satisfaction with treatment. Each item is rated by participant with a 3 point frequency scale:2=often, 1=sometimes, 0=never.Change in PETiT total score: total score at month 24 minus total score at randomization
Time Frame: Randomization to Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
units on scale | 1.2 (6.2) | 0.9 (6.0)

11. Secondary Outcome: Number of Relapses of Schizophrenia or Schizoaffective Disorder
Description: Relapse is defined as a hospital stay for psychiatric symptoms or a 2-point increase from baseline in the CGI severity score. CGI-S score ranges from 0-7 with 0 = Not Assessed, 1 = Normal, not at all and 7 = Among the most extremely ill subjects.
Time Frame: At Month 24
Population: as for outcome 4
Measure: Number; unit: Relapses
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 506 | 428
Relapses | 24 | 33

12. Secondary Outcome: Change in Simpson-Angus Scale (SAS) Total Score
Description: SAS total score is the sum of the 10 individual-item scores (range:0-40), with the score for each item ranging from 0 to 4, higher scores indicate greater severity of Parkinsonian symptoms. Change : total score at month 24 minus total score at randomization. Increase in Change of total score indicates an increase in extrapyramidal motor symptoms.
Time Frame: Randomization to Month 24
Population: The Safety analysis set included all randomized participants who received at least 1 dose of study medication
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 586 | 496
units on scale | -0.7 (2.1) | -0.4 (2.8)

13. Secondary Outcome: Change in Barnes Akathisia Rating Scale (BARS) Global Score
Description: BARS global score is the 4th individual-item score on the BARS scale, the Global Assessment of Akathisia, with the score ranging from 0 (no evidence of akathisia) to 5 (severe akathisia). Change : score at month 24 minus score at randomization. Increase in Change of BARS global score indicates an increase in akathisia.
Time Frame: Randomization to Month 24
Population: The Safety analysis set included all randomized participants who received at least 1 dose of study medication
Measure: Mean (Standard Deviation); unit: units of scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 586 | 496
units of scale | -0.1 (0.7) | 0.1 (0.8)

14. Secondary Outcome: Change in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: AIMS total score is the sum of the 10 individual-item scores(range:0-40), with the score for each item ranging from 0 to 4. Change : total score at month 24 minus total score at randomization. Increase in Change of total score indicates an increase in abnormal voluntary movements. The lower score means lower intensity of abnormal voluntary Movements. 0 is best, 4 is worst. Increase in Change of total score indicates an increase in abnormal voluntary Movements.
Time Frame: Randomization to Month 24
Population: The Safety analysis set included all randomized participants who received at least 1 dose of study medication
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 586 | 496
units on scale | -0.2 (2.5) | 0.1 (2.5)

15. Secondary Outcome: Number of Participants With Potential Extrapyramidal Symptoms (EPS)
Description: Number of participants with adverse events potentially associated with EPS collected by MedDRA Preferred Terms as akathisia, bradykinesia, drooling, dyskinesia, dystonia, extrapyramidal disorder, grimacing, muscle rigidity, parkinsonism, restlessness, tardive dyskinesia, tremor
Time Frame: From start of the study treatment to last dose plus 30 days
Population: The Safety analysis set included all randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Participants
Arm/Group | Quetiapine Fumarate | Risperidone
Number analyzed (Participants) | 586 | 496
Participants | 73 | 106

ADVERSE EVENTS:
Arm/Group | Quetiapine Fumarate | Risperidone
Serious Adverse Events (participants affected / at risk) | 151/596 | 114/502
Other Adverse Events (participants affected / at risk) | 476/596 | 368/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Quetiapine Fumarate (N=596) | Risperidone (N=502)
Anaemia (Blood and lymphatic system disorders) | 1/586 | 1/496
Angina Pectoris (Cardiac disorders) | 0/586 | 2/496
Cardiac Failure Congestive (Cardiac disorders) | 2/586 | 0/496
Arrhythmia (Cardiac disorders) | 0/586 | 1/496
Coronary Artery Disease (Cardiac disorders) | 0/586 | 1/496
Diastolic Dysfunction (Cardiac disorders) | 1/586 | 0/496
Myocardial Infarction (Cardiac disorders) | 1/586 | 0/496
Hyperparathyroidism (Endocrine disorders) | 0/586 | 1/496
Hypoparathyroidism (Endocrine disorders) | 0/586 | 1/496
Hypothyroidism (Endocrine disorders) | 0/586 | 1/496
Intestinal Ischaemia (Gastrointestinal disorders) | 0/586 | 1/496
Nausea (Gastrointestinal disorders) | 0/586 | 1/496
Pancreatic Insufficiency (Gastrointestinal disorders) | 0/586 | 1/496
Abdominal Discomfort (Gastrointestinal disorders) | 1/586 | 0/496
Anal Fistula (Gastrointestinal disorders) | 1/586 | 0/496
Colitis (Gastrointestinal disorders) | 1/586 | 0/496
Intestinal Obstruction (Gastrointestinal disorders) | 1/586 | 0/496
Pancreatitis (Gastrointestinal disorders) | 1/586 | 0/496
Pancreatitis Acute (Gastrointestinal disorders) | 1/586 | 0/496
Chest Pain (General disorders) | 2/586 | 0/496
Non-Cardiac Chest Pain (General disorders) | 2/586 | 0/496
Cholecystitis (Hepatobiliary disorders) | 0/586 | 1/496
Cholelithiasis (Hepatobiliary disorders) | 0/586 | 1/496
Cholecystitis Acute (Hepatobiliary disorders) | 1/586 | 0/496
Pneumonia (Infections and infestations) | 4/586 | 3/496
Appendicitis (Infections and infestations) | 1/586 | 1/496
Cellulitis (Infections and infestations) | 0/586 | 1/496
Conjunctivitis Bacterial (Infections and infestations) | 0/586 | 1/496
Diarrhoea Infectious (Infections and infestations) | 0/586 | 1/496
Diverticulitis (Infections and infestations) | 0/586 | 1/496
Gastroenteritis (Infections and infestations) | 1/586 | 1/496
Gastroenteritis Viral (Infections and infestations) | 0/586 | 1/496
Skin Infection (Infections and infestations) | 0/586 | 1/496
Urinary Tract Infection (Infections and infestations) | 1/586 | 1/496
Bronchitis (Infections and infestations) | 1/586 | 0/496
Localised Infection (Infections and infestations) | 1/586 | 0/496
Pilonidal Cyst (Infections and infestations) | 1/586 | 0/496
Postoperative Wound Infection (Infections and infestations) | 1/586 | 0/496
Sepsis (Infections and infestations) | 1/586 | 0/496
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1/586 | 3/496
Accidental Overdose (Injury, poisoning and procedural complications) | 2/586 | 2/496
Drug Toxicity (Injury, poisoning and procedural complications) | 0/586 | 2/496
Concussion (Injury, poisoning and procedural complications) | 0/586 | 1/496
Incisional Hernia (Injury, poisoning and procedural complications) | 0/586 | 1/496
Injury (Injury, poisoning and procedural complications) | 0/586 | 1/496
Intentional Overdose (Injury, poisoning and procedural complications) | 0/586 | 1/496
Joint Dislocation (Injury, poisoning and procedural complications) | 0/586 | 1/496
Laceration (Injury, poisoning and procedural complications) | 0/586 | 1/496
Multiple Drug Overdose Accidental (Injury, poisoning and procedural complications) | 0/586 | 1/496
Procedural Pain (Injury, poisoning and procedural complications) | 0/586 | 1/496
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0/586 | 1/496
Thermal Burn (Injury, poisoning and procedural complications) | 1/586 | 1/496
Ankle Fracture (Injury, poisoning and procedural complications) | 1/586 | 0/496
Contusion (Injury, poisoning and procedural complications) | 1/586 | 0/496
Respiratory Fume Inhalation Disorder (Injury, poisoning and procedural complications) | 1/586 | 0/496
Electrocardiogram Qt Prolonged (Injury, poisoning and procedural complications) | 1/586 | 0/496
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 1/586 | 0/496
Diabetes Mellitus (Metabolism and nutrition disorders) | 0/586 | 3/496
Dehydration (Metabolism and nutrition disorders) | 0/586 | 1/496
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0/586 | 1/496
Hypercalcaemia (Metabolism and nutrition disorders) | 0/586 | 1/496
Hypoglycaemia (Metabolism and nutrition disorders) | 0/586 | 1/496
Hypokalaemia (Metabolism and nutrition disorders) | 1/586 | 0/496
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0/586 | 1/496
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0/586 | 1/496
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0/586 | 1/496
Back Pain (Musculoskeletal and connective tissue disorders) | 1/586 | 0/496
Flank Pain (Musculoskeletal and connective tissue disorders) | 1/586 | 0/496
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1/586 | 0/496
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1/586 | 0/496
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1/586 | 0/496
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/586 | 1/496
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/586 | 0/496
Oesophageal Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/586 | 0/496
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/586 | 0/496
Dizziness (Nervous system disorders) | 0/586 | 2/496
Syncope (Nervous system disorders) | 2/586 | 0/496
Ataxia (Nervous system disorders) | 0/586 | 1/496
Convulsion (Nervous system disorders) | 0/586 | 1/496
Hemiparesis (Nervous system disorders) | 1/586 | 1/496
Migraine (Nervous system disorders) | 0/586 | 1/496
Transient Ischaemic Attack (Nervous system disorders) | 0/586 | 1/496
Dysarthria (Nervous system disorders) | 1/586 | 0/496
Multiple Sclerosis (Nervous system disorders) | 1/586 | 0/496
Presyncope (Nervous system disorders) | 1/586 | 0/496
Subarachnoid Haemorrhage (Nervous system disorders) | 1/586 | 0/496
Psychotic Disorder (Psychiatric disorders) | 38/586 | 19/496
Schizophrenia (Psychiatric disorders) | 25/586 | 20/496
Schizoaffective Disorder (Psychiatric disorders) | 19/586 | 14/496
Suicidal Ideation (Psychiatric disorders) | 12/586 | 12/496
Depression (Psychiatric disorders) | 13/586 | 8/496
Suicide Attempt (Psychiatric disorders) | 5/586 | 6/496
Schizophrenia, Paranoid Type (Psychiatric disorders) | 5/586 | 3/496
Anxiety (Psychiatric disorders) | 3/586 | 2/496
Aggression (Psychiatric disorders) | 2/586 | 0/496
Alcohol Abuse (Psychiatric disorders) | 2/586 | 0/496
Completed Suicide (Psychiatric disorders) | 2/586 | 1/496
Drug Abuse (Psychiatric disorders) | 2/586 | 0/496
Hallucination (Psychiatric disorders) | 2/586 | 0/496
Paranoia (Psychiatric disorders) | 2/586 | 0/496
Affective Disorder (Psychiatric disorders) | 0/586 | 1/496
Delusion (Psychiatric disorders) | 0/586 | 1/496
Homicidal Ideation (Psychiatric disorders) | 1/586 | 1/496
Major Depression (Psychiatric disorders) | 1/586 | 1/496
Acute Psychosis (Psychiatric disorders) | 1/586 | 0/496
Alcoholism (Psychiatric disorders) | 1/586 | 0/496
Catatonia (Psychiatric disorders) | 1/586 | 0/496
Drug Dependence (Psychiatric disorders) | 1/586 | 0/496
Flashback (Psychiatric disorders) | 1/586 | 0/496
Self Injurious Behaviour (Psychiatric disorders) | 1/586 | 0/496
Somatic Delusion (Psychiatric disorders) | 1/586 | 0/496
Substance Abuse (Psychiatric disorders) | 1/586 | 0/496
Suicidal Behaviour (Psychiatric disorders) | 1/586 | 0/496
Bladder Disorder (Renal and urinary disorders) | 0/586 | 1/496
Renal Failure Acute (Renal and urinary disorders) | 1/586 | 1/496
Breast Mass (Reproductive system and breast disorders) | 1/586 | 0/496
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4/586 | 0/496
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2/586 | 0/496
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/586 | 1/496
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0/586 | 1/496
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/586 | 1/496
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/586 | 1/496
Angioedema (Skin and subcutaneous tissue disorders) | 0/586 | 1/496
Substance Abuser (Vascular disorders) | 1/586 | 0/496
Hypertension (Vascular disorders) | 0/586 | 1/496
Malignant Hypertension (Vascular disorders) | 0/586 | 1/496
Arteriosclerosis (Vascular disorders) | 1/586 | 0/496
Hypotension (Vascular disorders) | 1/586 | 0/496
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Quetiapine Fumarate (N=596) | Risperidone (N=502)
Dry Mouth (Gastrointestinal disorders) | 78/586 | 39/496
Nausea (Gastrointestinal disorders) | 47/586 | 43/496
Constipation (Gastrointestinal disorders) | 45/586 | 28/496
Vomiting (Gastrointestinal disorders) | 21/586 | 36/496
Toothache (Gastrointestinal disorders) | 38/586 | 17/496
Diarrhoea (Gastrointestinal disorders) | 25/586 | 30/496
Fatigue (General disorders) | 60/586 | 46/496
Nasopharyngitis (Infections and infestations) | 54/586 | 50/496
Upper Respiratory Tract Infection (Infections and infestations) | 31/586 | 32/496
Weight Increased (Infections and infestations) | 69/586 | 41/496
Back Pain (Musculoskeletal and connective tissue disorders) | 42/586 | 30/496
Arthralgia (Musculoskeletal and connective tissue disorders) | 36/586 | 28/496
Somnolence (Nervous system disorders) | 169/586 | 64/496
Sedation (Nervous system disorders) | 135/586 | 54/496
Headache (Nervous system disorders) | 96/586 | 78/496
Dizziness (Nervous system disorders) | 84/586 | 49/496
Akathisia (Nervous system disorders) | 26/586 | 33/496
Tremor (Nervous system disorders) | 25/586 | 31/496
Extrapyramidal Disorder (Nervous system disorders) | 9/586 | 27/496
Insomnia (Psychiatric disorders) | 89/586 | 110/496
Anxiety (Psychiatric disorders) | 71/586 | 52/496
Depression (Psychiatric disorders) | 52/586 | 48/496
Cough (Respiratory, thoracic and mediastinal disorders) | 25/586 | 25/496

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate in good faith with AstraZeneca with regards to the contents and formation of any publication or disclosure to be made by the PI and to pay due consideration to the comments, views and opinions offered by AstraZeneca